CLINICAL TRIAL: NCT01972659
Title: Effects of Magnesium Sulphate on Sugammadex Reversal of Rocuronium Induced Blockade in Gynaecology Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Zehra Ipek ARSLAN, Assistant Professor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KOU 2012 KAEK 144
Record Dates: First submitted 2013-10-11; First posted 2013-10-30 (Estimated); Results first posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-01

CONDITIONS: Pre-eclampsia Aggravated
Keywords: sugammadex; rocuronium; magnesium; female
MeSH Terms: interventions — Sodium Chloride; Magnesium Sulfate; Magnesium; Sugammadex

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sugammadex and placebo (Active Comparator): sugammadex: 4 mg/kg iv bolus at the end of the surgery at a TOF count of 1 placebo: isotonic saline (%0.9 NaCl) 50 mg/kg iv bolus plus 15 mg/kg continuous infusion until the end of surgery
  Interventions: Drug: placebo; Drug: sugammadex
- sugammadex and magnesium sulphate (Experimental): sugammadex: 4 mg/kg iv bolus at the end of the surgery at a TOF count of 1 magnesium: 50 mg/kg iv bolus plus continuous infusion until the end of surgery
  Interventions: Drug: Magnesium Sulphate; Drug: sugammadex

INTERVENTIONS:
Drug: placebo — Active comparator 50 mg/kg iv bolus plus 15 mg/kg continuous infusion
  Other Names: %0.9 NaCl; isotonic saline
  Arms: sugammadex and placebo
Drug: Magnesium Sulphate — Experimental :
  50 mg/kg bolus plus 15 mg/kg continuous infusion
  Other Names: magnesium
  Arms: sugammadex and magnesium sulphate
Drug: sugammadex — 4 mg/kg iv bolus at the end of the surgery
  Other Names: bridion

SUMMARY:
Background: The aim of this prospective study was to evaluate the effect of magnesium on the reversal of rocuronium-induced neuromuscular block by sugammadex.

Methods: Eighty patients, aged 18 to 60 years, American Society of Anesthesiologists I-II, undergoing elective gynecological surgery were enrolled. Anaesthesia was induced with propofol and fentanyl and was maintained with 60% nitrous oxide and Oxygen in sevoflurane. The magnesium group received 50 milligram/kilogram (mg/kg) Magnesium intravenous (iv) as a bolus and 15 mg/kg/hour by continuous infusion until the completion of surgery. The placebo group received the equivalent volume of isotonic saline. For intubation, 0.6 mg/kg rocuronium was administered and 0.1 mg/kg was added when Train of four (TOF) counts reached 1 or more during the procedure. At the end of the surgery at a TOF count of 1, 4 mg/kg sugammadex iv was administered. Patients were observed until a TOF ratio of 0.9 was achieved. Patient-controlled analgesia with intravenous morphine was used postoperatively.

DETAILED DESCRIPTION:
Inclusion criteria:

* American Society of Anesthesiologists physical status I or II
* 18-60 years of age
* undergoing elective gynecological surgery
* requiring endotracheal intubation

Exclusion criteria:

* Patients who had body mass index > 35
* gastroesophageal reflux
* a history of allergy
* used medication known to interact with the drugs being used in this trial
* who experienced expected or unexpected difficulty during intubation or ventilation
* had neuromuscular disease
* hepatic or renal insufficiency
* pregnant
* were American Society of Anesthesiologists III or IV
* had a family history of malignant hyperthermia
* detection if low or high control plasma magnesium levels

ELIGIBILITY:
Inclusion Criteria:

* female patients
* American Society of Anesthesiologists (ASA) physical status I or II
* 18-60 years of age who were undergoing elective gynecological surgery
* requiring endotracheal intubation were enrolled in this prospective study.

Exclusion Criteria:

* Patients who had body mass index > 35
* gastroesophageal reflux
* a history of allergy
* used medication known to interact with the drugs being used in this trial
* who experienced expected or unexpected difficulty during intubation or ventilation
* had neuromuscular disease
* hepatic or renal insufficiency
* were pregnant
* had a family history of malignant hyperthermia
* detection if low or high control plasma magnesium levels

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zehra I. ARSLAN, Asst. Prof., Principal Investigator — Anesthesiology and Reanimation
Locations (1):
- Kocaeli University Hospital, Kocaeli, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugammadex and Magnesium Sulphate: sugammadex: 4 mg/kg iv bolus at the end of the surgery at a TOF count of 1 magnesium: 50 mg/kg iv bolus plus continuous infusion until the end of surgery
  Magnesium Sulphate: Experimental :
  50 mg/kg bolus plus 15 mg/kg continuous infusion
  sugammadex: 4 mg/kg iv bolus at the end of the surgery
Period: Overall Study
Arm/Group | Sugammadex and Placebo | Sugammadex and Magnesium Sulphate
Started | 40 | 40
Completed | 36 | 37
Not Completed | 4 | 3
Not completed — Protocol Violation | 2 | 2
Not completed — problems realted to acceleromyograph | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex and Placebo | Sugammadex and Magnesium Sulphate | Total
Number analyzed (Participants) | 36 | 37 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (10.3) | 39.4 (10.6) | 40.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 37 | 73
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: TOF 0.9 Achieving Time
Time Frame: end of the surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex and Placebo | Sugammadex and Magnesium Sulphate
Number analyzed (Participants) | 36 | 37
minutes | 1.6 (0.6) | 2.1 (0.9)

2. Secondary Outcome: Rocuronium Onset Time
Time Frame: during the surgery
Reporting Status: Not Posted

3. Secondary Outcome: Rocuronium Supplementation
Time Frame: during surgery
Reporting Status: Not Posted

4. Secondary Outcome: Postoperative Morphine Consumption
Time Frame: after 12 hour surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Sugammadex and Placebo | Sugammadex and Magnesium Sulphate
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No